CLINICAL TRIAL: NCT05913479
Title: HYDRAGYNE (MUCG234) - Evaluation of the Efficacy and Safety of Mucogye® Gel as a Moisturizer
Brief Title: Evaluation of the Efficacy and Safety of Mucogye® Gel as a Moisturizer
Acronym: HYDRAGYNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biocodex (Industry)
Collaborators: Voisin Consulting Life Science (VCLS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MUCG234; 2022-A02088-35 (Other: ID-RCB)
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Vaginal Dryness

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter (France), open label without comparator study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mucogyne treatment (Experimental): 3 planned visits for each eligible patient:
  * Screening/Baseline visit: V0 at Day 0. Patient receive a box of Mucogyne Gel.
  * Phone call: V1 phone call at Day 10 ± 3
  * End-of-study visit: V2 at Day 35 ± 3
  Interventions: Device: Mucogyne Gel

INTERVENTIONS:
Device: Mucogyne Gel — At inclusion visit (V0), the Investigator will ask the subject to apply MUCOGYNE® Gel as described in the Instructions For Use, i.e., internally, one application 2 to 3 times a week until symptoms improve during 5 weeks (D35 +/- 3)

SUMMARY:
The aim of this post-Market Clinical Follow-up (PMCF) study for a class IIb medical device is to confirm th efficacy and safety of Mucogyne Gel as a moisturizer in women with vaginal dryness irrespective of the cause; when used in accordance with its approved labelling.

ELIGIBILITY:
Inclusion Criteria:

Women with the following conditions:

* ≥ 18 years of age at inclusion with vaginal dryness, irrespective of the cause (which may or may not be accompanied by irritation of the vulva, discomfort, or itchiness).
* Having a Vaginal Health Index Score (VHIS) <15 associated to pain and/or dyspareunia feeling.
* Subject agrees to not use any lubricant, local estrogens, or other vaginal product during the study.
* Subject agrees to not modify their intimate hygiene products.
* Able to understand and sign the informed consent form for study enrolment.
* Subject able to comply with study requirements, as defined in the protocol.
* Subject affiliated to a health social security system.

Exclusion Criteria:

Women with the following conditions:

* General:

  * Pregnancy (subject of childbearing potential must not be pregnant and must agree to avoid pregnancy during the study by using an effective birth control method from at least one month before D0 (V0) and throughout the duration of the study).
  * Participating at the same time in another interventional trial within the four previous weeks and during the study period, being in an exclusion period for a previous study.
  * Deprived of freedom by administrative or legal decision or under guardianship.
  * Subject in a social or sanitary establishment.
  * Subject suspected to be non-compliant according to the investigator's judgment.
  * Subject in an emergency situation.
* Linked to subject's status:

  * Known hypersensitivity to one of MUCOGYNE® Gel components.
  * Subject with a known vaginal pathology (clinical diagnosis only) other than vaginal dryness/atrophy.
* Linked to previous or ongoing treatments:

  * Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk.
  * Subject suffering from systemic diseases and/or using concurrent therapy that may interfere with the evaluation of the study results.
  * Subject undergoing a topical treatment on the test area or a systemic treatment: corticosteroids during the 2 previous weeks and during the study; retinoids and/or immunosuppressors during the 1,5 previous months and during the study; subject having started or changed her oral contraceptive or any other hormonal treatment during the one previous month.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the efficacy of MUCOGYNE® Gel intra vaginal applications on subjects' vaginal dryness irrespective of the cause over a 35-day period of use. | Day 0 to Day 35 +/- 3
  Primary efficacy criterion: Clinical scoring, by the investigator, of the Vaginal Health Index Score (VHIS), including evaluation of elasticity, fluid volume, pH, epithelial integrity, and moisture.

SECONDARY OUTCOMES:
Assessment of the local performance of MUCOGYNE® Gel in reducing vulva irritation | Day 0 to Day 35 +/- 3
  Secondary efficacy criteria
  - Auto-evaluation, by the subjects, of pain and/or dyspareunia on Visual Analogical Scales (VAS) from 0 to 10
Assessment of the local performance of MUCOGYNE® Gel in reducing vulvo-vaginal dryness | Day 0 to Day 35 +/- 3
  Secondary efficacy criteria
  - Clinical scoring of vulvo-vaginal dryness by the Investigator on a Visual Analogical Scale from 0 to 10
Assessment by investigator of changes in patient's clinical status | Day 0 to Day 35 +/- 3
  Secondary efficacy criteria
  - Completion of the CGI-I (Clinical Global Impressions-Improvement) by the Investigator.
Assessment of changes in patient's clinical status | Day 0 to Day 35 +/- 3
  Secondary efficacy criteria
  - Completion of the Patients' Global Impression of Change (PGIC) Scale to assess the changes perceived by the patient following the treatment taken.
Assessment of the patient's satisfaction | Day 0 to Day 35 +/- 3
  Secondary efficacy criteria
  - Completion of the intra vaginal treatment satisfaction questionnaire (Likert questionnaire) to assess the level of satisfaction of the treatment on the vaginal symptoms.
Assessment of the patient's sexual function | Day 0 to Day 35 +/- 3
  Secondary efficacy criteria
  - Completion of the self-reported FSFI (Female Sexual Function Index) to investigate sexual function (for women having sexual relations).

CONTACTS AND LOCATIONS:
Overall Officials: Oana BERNARD, MD, Study Director — Chief Scientific officer
Locations (4):
- France (4):
  - Dr Paul Lefevre's medical office, Caen
  - Dr Thierry KELLER's medical office, Colmar
  - Dr Christiane ARMAND's medical office, Écully
  - Sihame MOKHBAT's office, Paris